CLINICAL TRIAL: NCT03177941
Title: Validation of Mobile Technologies for Clinical Assessment, Monitoring, and Intervention (SBIR Topic 342, Direct to Phase II- Vignet, Inc.)
Brief Title: Teaching Skin Self-Examination to First-degree Relatives of Melanoma Patients Using Mobile App Technology
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The company decided not to enroll subjects. The app was never developed.
Sponsor: Northwestern University (Other)
Collaborators: Vibrent Health (Industry); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, June Robinson, MD, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STU00204232
Record Dates: First submitted 2017-06-02; First posted 2017-06-06 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Melanoma
Keywords: Melanoma; Skin Self-Examination; First-degree Relative; Mobile Application
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Intervention Model Description: 2 Group Random Clinical Trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Skin Self-Examination (Experimental): Melanoma patients (n=300) and their first-degree relatives (n=300) that are between 16-70 years old will participate in the study. Participants will be randomized to receive the intervention or the control group. Participants randomized to the control group will have access to the app later.
  Assigned Interventions Behavioral: Skin self-examination structure training First-degree relatives download a mobile application onto their smart phone (n=150). This is the skin self-examination training intervention used in the original RCT (MoleScore). Participants will perform a Skin Self-Examination with partner assistance each month during the study. Participants will take a picture of one of their moles using their smart phone and upload to the application one image of a mole/freckle with a decision about their mole/freckle.
  Interventions: Other: Eviderma Smart Phone Teledermatology Application (Eviderma)
- Active Control (Active Comparator): Participants (n=150) will complete web-based surveys at baseline and 4-months. Control participants do not initially receive training; however, after completing the 4-month survey they will be given access to the training.
  Assigned Interventions
  Behavioral: Skin self-examination structured training Training will be provided via a mobile application. After completing the 4-month survey, the control participants may request the link to download the application.
  Interventions: Other: Eviderma Smart Phone Teledermatology Application (Eviderma)

INTERVENTIONS:
Other: Eviderma Smart Phone Teledermatology Application (Eviderma) — First-degree relatives download a mobile application onto their smart phone (n=150). This is the skin self-examination training intervention used in the original RCT (MoleScore). Participants will perform a Skin Self-Examination with partner assistance each month during the study. Participants will take a picture of one of their moles using their smart phone and upload to the application one image of a mole/freckle with a decision about their mole/freckle.

SUMMARY:
The proposed study builds upon the success of our research program (STU00017005: Interventions to teach melanoma patients skin self-examination and the continuation STU0201983) designed to increase early detection of melanomas before they metastasize. This study seeks to expand the use of our efficacious skin self-examination (SSE) training program to first-degree relatives with automated support with reminders and the dermatologist coaching about pictures of moles submitted by user. In 2015 there are more than 1 million living melanoma patients in the United States (US), and almost 500,000 were age 40-60 years. If each melanoma patient has 2.79 first-degree relatives (children, and siblings of melanoma patients), then there are 2.79 million first-degree relatives and 1 million melanoma patients or 3.79 million people at-risk to develop melanoma, who are predominantly non-Hispanic White. A first-degree relative (FDR) is the parent, sibling or child of a melanoma patient. In 2015, approximately 73,870 individuals in the US will be diagnosed with invasive melanoma and about 9,940 will die from the disease. People with a history of melanoma have 10 times greater risk of developing a second new melanoma relative to the general population. A first-degree relative of a melanoma patient (parent, child, sibling) has an 8 times greater chance of developing melanoma. Early detection with surgical excision at an early stage when treatment is usually more effective is the only proven curative strategy. Thus, enhanced surveillance for melanoma patients and screening for their first-degree relatives, who have the same skin type (skin that easily sunburns) and melanoma-risk habits (sunny vacations) as the melanoma survivor, has the potential to detect melanomas in the early stages where treatment prognosis is optimal. Indeed, several societies recommend routine screening by a physician for persons with a family history of melanoma.

DETAILED DESCRIPTION:
The melanoma diagnosis represents a patchwork of transitions for the family with the opportunity to promote early detection in the first-degree relatives of melanoma patients. While family communication is a promising way to promote risk awareness and provide skills training in skin self-examination (SSE), knowing about a family member with a history of melanoma is no guarantee that a relative will accept their risk or act to minimize their risk by performing SSE. Indeed performance of SSE by people at-risk to develop melanoma ranges from 39% to 50%. Family separation by distance can now be overcome with technology (Skype, Facetime), but support for melanoma patients, who frame the risk of developing melanoma for their relatives, does not exist. The melanoma patient needs to be a) confident in their ability to communicate with at-risk relatives, b) able to reassure their loved one(s) that they can learn to do a skin check and perform it well, and c) supported in their decisions about pigmented lesions (moles) by ready access to a physician. The tools to learn how to check for melanoma with the assistance of a partner to see locations that are difficult for a person to see on their own body, e.g. the back and tops of the ears have been developed and validated by Robinson et al. Now, we will use of informatics technology of the proven physician-to-physician consultation of the Vibrent Mobile Telederm system to provide first-degree relatives of melanoma patients with education about their risk of developing melanoma and the importance of early detection, teach the skills to perform SSE, provide diaries for home use and access to a dermatologist. The first-degree relative will download the Eviderma Smart Phone Teledermatology Application (Eviderma), learn how to perform SSE, and self-report their adherence to their care plan by reporting their SSE results, and send the dermatologist a picture of one pigmented lesion (mole) each month with scores of the features and a decision about whether it is concerning, and the dermatologist will recommend next steps. The first-degree relative will benefit from automated self-service supported via tailored content and evidence-based health literacy and educational content. This program gives the first-degree relative of the melanoma patient the right information at the right time to learn the skills needed to detect concerning lesions without unnecessary visits to the doctor, thus, saving cost.

The study aims are as follows:

1. To expand the uptake of an efficacious evidence-based SSE training program to first-degree relatives with the Eviderma program.

   * Eviderma develops materials for the first-degree relatives of melanoma patients, and improves their education and awareness of the risk of developing melanoma.
   * Assess engagement of first-degree relatives within the Eviderma program.
2. To assess the efficacy of the Eviderma program for melanoma patients' first-degree relatives.

   * A randomized controlled trial with the first-degree relatives of melanoma patients diagnosed with Stage 0-IIIA within the last five years
   * Assess change from baseline to 4 months in: a) knowledge about melanoma b) perception of risk of developing melanoma and importance of early detection b) SSE skills c) SSE performance, d) physician visits
3. To examine for whom the Eviderma program works best/least by assessing baseline perceived risk, importance of melanoma and its early detection, SSE self-efficacy and sex moderate SSE performance.
4. Assess health care expenditures of first-degree relatives using the Eviderma program in comparison with controls for the cost of visits with the primary care physician and dermatologist, including biopsy of lesions and their pathology

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria for Melanoma Patient:

  * Melanoma patient with Stage 0-IIIA diagnosed within the last 5 years
  * At least 2 months post-surgical treatment
  * Age 18-70 years old
  * Has Internet access
  * Owns and can use a smartphone
  * Has an adult (18-70 years old) first-degree relative (sibling, parent, child)
  * Willing to recruit a first-degree relative to be educated in SSE
  * If the melanoma patient is selected to participate as a skin check partner by their first-degree relative, then they may serve as a skin check partner over the duration of the 4 months; however, no data is collected from skin check partners.

Inclusion Criteria for First-degree Relative:

* Have a first-degree relative who is melanoma patient with Stage 0-IIIA diagnosed within the last five years
* No personal history of melanoma
* Age 18-70 years old
* Teen child 16 to 17 years of age.
* Owns and can use a smartphone that can take close-up pictures of moles and can upload pictures of moles to the HIPPA secure website
* Has Internet access
* Willing to participate in two online assessments with an optional third survey if the person finds a clinically concerning mole and has an appointment with a primary care physician or a dermatologist to evaluate the clinically concerning mole, and receive reminders via the mobile device

Exclusion Criteria:

- Exclusion Criteria for Melanoma Patient:

• Subjects overburdened with other co-morbid diseases (e.g. chronic immunosuppression from organ transplantation) or medical treatments (e.g. chemotherapy)

Exclusion Criteria for First-degree Relative:

* Subjects overburdened with other co-morbid diseases (e.g. chronic immunosuppression from organ transplantation) or medical treatments (e.g. chemotherapy)
* Do not own a smartphone

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Performance of skin-self examination | 4-months
  The first-degree relative and their skin check partner check about 5 moles/ freckles monthly, and upload a photograph of one mole with a decision about whether the mole is benign, needs to be watched for change, or may be malignant and they need to see a doctor.

SECONDARY OUTCOMES:
Engage a partner in helping to check hard to see locations. | 4-months
  Self- reported responses to survey

CONTACTS AND LOCATIONS:
Overall Officials: June K. Robinson, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine Department of Dermatology, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Publish results

REFERENCES:
- [Background] Robinson JK, Gaber R, Hultgren B, Eilers S, Blatt H, Stapleton J, Mallett K, Turrisi R, Duffecy J, Begale M, Martini M, Bilimoria K, Wayne J. Skin self-examination education for early detection of melanoma: a randomized controlled trial of Internet, workbook, and in-person interventions. J Med Internet Res. 2014 Jan 13;16(1):e7. doi: 10.2196/jmir.2883. PMID 24418949